CLINICAL TRIAL: NCT01111513
Title: The Influence of the Femoral Nerve Block on the Quadriceps Strength After Total Knee Replacement
Brief Title: The Influence of the Femoral Nerve Block on Quadriceps Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital de l'Enfant-Jesus (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEJ-413
Record Dates: First submitted 2010-04-21; First posted 2010-04-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Total Knee Arthroplasty
Keywords: knee surgery; total knee arthroplasty; total knee replacement; ropivacaine; femoral nerve block
MeSH Terms: interventions — Ropivacaine; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous femoral block (Active Comparator): Patients receive a continuous femoral block for 48 hours and they have patient controlled analgesics.
  Interventions: Drug: 48-hour ropivacaine infusions
- Single dose femoral block (Active Comparator): Patients receive a single dose femoral block and have patient controlled analgesics.
  Interventions: Drug: Single dose ropivacaine
- Patient controlled analgesics (Active Comparator): Patients do not receive a femoral block. They only have patient controlled analgesics.
  Interventions: Drug: Patient controlled analgesics

INTERVENTIONS:
Drug: 48-hour ropivacaine infusions — Patients receive 20 ml of ropivacaine 0.5 % pre-operation through femoral block catheter, followed by ropivacaine infusions from 0.1 % to 0.1 ml/kg/hour for 48 hours.
  Other Names: ropivacaine; femoral block
  Arms: Continuous femoral block
Drug: Single dose ropivacaine — Patients receive 20 ml of ropivacaine 0.5% pre-operation
  Other Names: ropivacaine
  Arms: Single dose femoral block
Drug: Patient controlled analgesics — Patient controlled analgesics alone, no femoral block
  Other Names: analgesics
  Arms: Patient controlled analgesics

SUMMARY:
Total knee replacement is a frequent procedure in Québec's hospitals and the muscular strength of the quadriceps is the best indicator of the patient's functional recovery post surgery. Thus, the importance of the patient's recovery leads to the evaluation of the influence of the femoral nerve block on the muscle strength.

The purpose of the study is to compare the short term and long term recuperation of the quadriceps' motor strength of after a total knee arthroplasty using different types of analgesics such as the continuous femoral nerve block, the single dose femoral nerve block and the systemic analgesic, a patient controlled analgesic pump.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* men or women needing an elective total knee replacement surgery

Exclusion Criteria:

* unicompartmental arthroplasty
* revision surgery for knee arthroplasty
* previous surgery on same knee
* previous fracture of femur/patella with functional after-effects
* allergies or contraindication to any medication used during study or to local anaesthesia technique
* preexisting neurological deficit
* severe anomaly of intracardiac conduction
* previous vascular surgery near the site of introduction of the catheter
* pregnancy or breastfeeding
* ASA IV or V14 class
* Men or women > 18 years old unfit to consent
* < 18 years old
* Refusal to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-11; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Quadriceps strength measurement with Cybex machine | 6 weeks after surgery
  Evidence of the influence of the different types of analgesics on the strength of the quadriceps post surgery. Quadriceps strength will be evaluated in open chain and closed chain with the help of the Cybex machine.
Quadriceps strength measurement with Cybex machine | 6 months after surgery
  Evidence of the influence of the different types of analgesics on the strength of the quadriceps post surgery. Quadriceps strength will be evaluated in open chain and closed chain with the help of the Cybex machine.
Quadriceps strength measurements with Cybex machine | 12 months after surgery
  Evidence of the influence of the different types of analgesics on the strength of the quadriceps post surgery. Quadriceps strength will be evaluated in open chain and closed chain with the help of the Cybex machine.

SECONDARY OUTCOMES:
Overall functional recovery | 6 weeks after surgery
  The overall functional recovery of the patient will be evaluated considering the analgesic type using SF-36 and WOMAC questionnaires.
Pain score on Visual Analog Scale (VAS) | every 6 hour for the 48 hours following surgery
  Evaluation of the effectiveness of the analgesics on pain with VAS .
Hospital stay length | 4 to 7 days after surgery
  Evaluation of the hospital stay length after total knee replacement taking into account the different types of analgesics.
Overall functional recovery | 6 months after surgery
  The overall functional recovery of the patient will be evaluated considering the analgesic type using SF-36 and WOMAC questionnaires.
Overall functional recovery | 12 months after surgery
  The overall functional recovery of the patient will be evaluated considering the analgesic type using SF-36 and WOMAC questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital Enfant-Jésus; Michèle Angers, PhD, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada